CLINICAL TRIAL: NCT00081575
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Comparative Study Of The Efficacy And Safety Of Intravenous Tigecycline Vs Intravenous Levofloxacin To Treat Subjects Hospitalized With Community-Acquired Pneumonia
Brief Title: Study Comparing Tigecycline vs. Levofloxacin in Subjects Hospitalized With Community-Acquired Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 3074A1-313
Record Dates: First submitted 2004-04-15; First posted 2004-04-19 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Community-Acquired Infections; Bacterial Pneumonia; Cross Infection
Keywords: Bacterial Pneumonia
MeSH Terms: conditions — Community-Acquired Infections; Pneumonia, Bacterial; Cross Infection | interventions — Tigecycline; Levofloxacin

INTERVENTIONS:
Drug: Tigecycline
Drug: Levofloxacin

SUMMARY:
To compare the efficacy and safety of IV tigecycline to IV levofloxacin in the treatment of subjects with CAP requiring hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 18 years of age and in Bulgaria only ≤ 70 years of age
* Subjects hospitalized with CAP with a severity that requires IV antibiotic treatment for at least 7 days
* The presence of fever (within 24 hours before randomization)

Exclusion Criteria:

* Any concomitant condition that, in the opinion of the investigator, would preclude an evaluation of a response or make it unlikely that the contemplated course of therapy could be completed (eg, life expectancy <30 days).
* Hospitalization within 14 days before the onset of symptoms.
* Residence in a long-term care facility or nursing home ≥14 days before the onset of symptoms.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2004-01; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Clinical response in the clinically evaluable population and the clinical modified intent-to-treat population at the TOC visit.
Determine whether tigecycline is noninferior to levofloxacin.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Ramirez JA, Cooper AC, Wiemken T, Gardiner D, Babinchak T; 308 Study Group. Switch therapy in hospitalized patients with community-acquired pneumonia: tigecycline vs. levofloxacin. BMC Infect Dis. 2012 Jul 19;12:159. doi: 10.1186/1471-2334-12-159. PMID 22812672
- [Derived] Tanaseanu C, Milutinovic S, Calistru PI, Strausz J, Zolubas M, Chernyak V, Dartois N, Castaing N, Gandjini H, Cooper CA; 313 Study Group. Efficacy and safety of tigecycline versus levofloxacin for community-acquired pneumonia. BMC Pulm Med. 2009 Sep 9;9:44. doi: 10.1186/1471-2466-9-44. PMID 19740418
- [Derived] Dartois N, Castaing N, Gandjini H, Cooper A; Tigecycline 313 Study Group. Tigecycline versus levofloxacin for the treatment of community-acquired pneumonia: European experience. J Chemother. 2008 Oct;20 Suppl 1:28-35. doi: 10.1179/joc.2008.20.Supplement-1.28. PMID 19036672
- [Derived] Tanaseanu C, Bergallo C, Teglia O, Jasovich A, Oliva ME, Dukart G, Dartois N, Cooper CA, Gandjini H, Mallick R; 308 Study Group; 313 Study Group. Integrated results of 2 phase 3 studies comparing tigecycline and levofloxacin in community-acquired pneumonia. Diagn Microbiol Infect Dis. 2008 Jul;61(3):329-38. doi: 10.1016/j.diagmicrobio.2008.04.009. Epub 2008 May 27. PMID 18508226